CLINICAL TRIAL: NCT03833960
Title: Impact of Sentinel Lymph Node Biopsy After Neoadjuvant Treatment on Locoregional Control of Disease in Initially Node Positive Breast Cancer Patients
Brief Title: SLNB After Neoadjuvant Treatment in Node Positive Patients
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Ana Car Peterko, general surgeon, Clinical Hospital Center Rijeka
Other Study IDs: SLNBvsALND
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Sentinel Lymph Node Biopsy; Locoregional Neoplasm Recurrence; Progression, Disease
Keywords: breast cancer; Sentinel Lymph Node Biopsy; Neoadjuvant Chemotherapy; locoregional recurrence; distant recurrence
MeSH Terms: conditions — Neoplasm Recurrence, Local; Disease Progression; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1-cN0/pN0: Patients with initially clinically negative axilla (cN0), submitted to neoadjuvant treatment, followed by surgical procedure within ALND or SLNB was done, and the final pathological report was ypN0.
- 2-cN+/pN0: Patients with initially clinically involved axilla (cN1-2), submitted to neoadjuvant treatment, followed by surgical procedure within ALND or SLNB was done, and the final pathological report was complete axillary remission (ypN0).
- 3-cN0/pN+: Patients with initially clinically negative axilla (cN0), submitted to neoadjuvant treatment, followed by surgical procedure within SLNB was done, followed by ALND because of positive pathological report of sentinel node(s).
- 4-cN+/pN+: Patients with initially clinically positive axilla (cN1-3) submitted to neoadjuvant treatment, followed by surgical procedure within ALND was done and the final pathological report was ypN1-3.

SUMMARY:
From May 2016 till May 2018 all breast cancer patients with operable disease submitted to surgery after neoadjuvant treatment would be divided in four groups considering initially clinical axillary stage, axillary procedure that was done, axillary response to preoperative systemic treatment and pathological axillary stage.

In first postoperative year all patients will be monitored for appearance of locoregional and distant recurrence.

DETAILED DESCRIPTION:
From May 2017 SLNB after neoadjuvant treatment was introduced in clinical practice for breast cancer patients presenting initially with involved axilla but shifted to clinically negative followed neoadjuvant treatment. This retrospective analysis is designed for period of one year before and one year later to compare the clinical outcomes for this patients in the setting where ALND was performed to the setting where SLNB was performed.

The main hypothesis was to establish that SLNB after neoadjuvant treatment, in initially node positive breast cancer patients that achieve complete clinical remission following neoadjuvant treatment, is reliable alternative to ALND in maintenance of locoregional control of disease.

For the purpose of this trial four groups were created and the results would be compared among them. In first postoperative year patients were monitored for the appearance of locoregional and distant recurrence.

Data were collected individually for each patient and recorded in register. All data are available to all members of investigation team, members of Ethic Committee and statistician.

Data collected in this trial would be used for publication.

ELIGIBILITY:
Inclusion Criteria:

* operable breast cancer submitted to neoadjuvant treatment in CHC Rijeka, followed by surgery in period from May 2016 till May 2018

Exclusion Criteria:

* T4 stage
* inflammatory breast cancer
* M1 stage at the time of diagnose
* bilateral disease
* multicentric disease
* unavailable complete required data

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Groups are formed from breast cancer patients with operable disease and involved axillary nodes, submitted to preoperative systemic treatment followed by surgical procedure in CHC Rijeka in period from May 2016 till May 2018
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Regional recurrence | 3 years
  All patients would be monitored in postoperative period of minimally one year for the appearance of locoregional recurrence. Results will be compared among all node negative patients (group 1 and 2) submitted to SLNB vs. ALND, and among group 2 patients only (ALND vs. SLNB).
Distant recurrence (progression) | 3 years
  All patients would be monitored in postoperative period of minimally one year for appearance of distant recurrence (disease progression). Results will be compared among patients from groups 2 and 4 and among group 2 patients only (ALND vs SLNB).

OTHER OUTCOMES:
Postoperative complications | 3 years
  To compare prolonged axillary serous secretion and arm lymphedema among patients submitted to ALND and SLNB.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Car Peterko, Principal Investigator — Clinical Hospital Center Rijeka